CLINICAL TRIAL: NCT03474302
Title: Program for African American Cognition & Exercise
Acronym: PAACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: BrightFocus Foundation (Other)
Responsible Party: Principal Investigator, Robert L. Newton, Jr., Associate Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-022
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Aging
Keywords: African American; Aging; Physical activity; Cognition
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The randomized controlled trial will assign insufficiently active African American adults aged 65-85 to an intervention or successful aging control group
Who Masked: Outcomes Assessor
Masking Description: Assessors will not know the group randomization of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (Experimental): The intervention will be a 12-week community-based physical activity promotion program
  Interventions: Behavioral: Physical Activity
- Successful Aging (Active Comparator): Those randomized to the successful aging group will receive health information pertinent to African Americans over the 12 weeks
  Interventions: Other: Successful Aging

INTERVENTIONS:
Behavioral: Physical Activity — Aerobic, strength training, balance, flexibility
  Arms: Physical Activity
Other: Successful Aging — Healthy aging education
  Arms: Successful Aging

SUMMARY:
The study is designed to develop and evaluate a physical activity promotion program among elderly African Americans with a long-term goal of reducing risk of Alzheimer's disease. The motivation for this study is that previous exercise interventions have improved cognitive function in older adults with and without cognitive impairments, but these studies were largely conducted without substantial African American representation. Due to genetic and environmental differences between African American and other populations, it is unclear whether positive findings from previous interventions will translate to African American individuals. Investigators hypothesize that a community-based physical activity intervention will a) be tailored to African American adults, b) increase daily amounts of physical activity, and c) improve cognitive function in sedentary older African American adults.

DETAILED DESCRIPTION:
Investigators will randomize 56 older African American adults into 1) a physical activity intervention specifically tailored to older African American or 2) a successful aging group. The 12-week physical activity intervention will consist of group based exercise sessions at a community facility and the successful aging groups will occur at Pennington Biomedical. Cognitive functioning and blood markers of circulating neurotrophic factors will be assessed to determine the brain effects of physical activity in this understudied population.

Specific Aim 1: To tailor a physical activity promotion intervention to community-dwelling African American elderly adults. Investigators will use focus groups to gather information needed to tailor a physical activity program to elderly African Americans.

Specific Aim 2: To determine if a physical activity promotion intervention in African American adults is effective in modifying physical activity and biological markers.

Specific Aim 3: To determine if a physical activity promotion intervention in African American adults benefits cognition and brain health. Change over the course of the intervention will be assessed in key AD related cognitive domains (memory, executive function, and processing speed).

Collecting this data sets the stage for the definitive study of exercise benefits on measures of amyloid, tau, inflammation, brain metabolism, and other AD-relevant pathways in elderly African Americans, which could in turn increase understanding of neurobiological mechanisms and optimal physical activity recommendations for elderly African Americans.

ELIGIBILITY:
Inclusion Criteria:

1. 65 - 85 years of age
2. African American
3. sedentary or insufficiently active
4. not cognitively impaired
5. physically capable of exercise
6. willing to accept randomization
7. willing to attend group sessions
8. willing to live in the study area for the next 6 months
9. willing to allow researchers to use data for research purposes after study participation is completed
10. free of conditions that would make regular exercise unsafe as deemed by the medical investigator

Exclusion Criteria:

1. unable or unwilling to give informed consent or accept randomization in either study group
2. are cognitively impaired (MMSE score of ≤ 26)
3. are unable to complete physical activity requirements (SPPB ≤ 3, complete 2 minute walk without sitting or resting against a surface)
4. are too active (steps per day > 50th percentile for age and gender)
5. have uncontrolled hypertension (systolic blood pressure > 200 mmHg and/or diastolic blood pressure > 110 mmHg).
6. gave had a hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
7. have had a myocardial infarction, major heart surgery (i.e., valve replacement or bypass surgery), stroke, deep vein thrombosis or pulmonary embolus in the past 6 months
8. are undergoing physical therapy or cardiopulmonary rehabilitation
9. are currently enrolled in another randomized trial involving lifestyle or pharmaceutical interventions
10. have another member of the household that is a participant in PAACE
11. have plans to relocate out of the study area within the next 6 months
12. have uncontrolled diabetes that in the judgment of the MI may interfere with study participation
13. have other medical, psychiatric, or behavioral factors that in the judgment of the Principal or Medical Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in steps. | 7-day period
  Steps will be measured by the abtigraph WGT3X+ accelerometer.

SECONDARY OUTCOMES:
Change in dementia screening. | Week 0 and Week 12
  The Mini-Mental State Examination (MMSE) is a 30-item measure of cognitive function. Scores range from 0-30, higher scores represent better global cognitive functioning.
Change in cognition. | Week 0 and Week 12
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a brief, individually administered battery to measure cognitive decline or improvement. Four subtests of the full battery of 12 subtests used to assess immediate memory (List Learning and Story Memory), as well as language capacities (i.e., Picture Naming and Semantic Fluency). T-scores are derived, higher scores represent better functioning.
Change in quality of life. | Week 0 and Week 12
  The Health Related Quality of Life questionnaire consists of 27 questions.
Change in health care utilization. | Week 0 and Week 12
  The Health Care Utilization questionnaire consists of 12 questions. Participants report utilization of various health care avenues.
Change in depressive symptoms. | Week 0 and Week 12
  The Geriatric Depression Scale (GDS) measures depressive symptoms specifically in an elderly population. Total scores range from 0 (no depressive symptoms) to 15 (indicative of depression).
Change in resilience. | Week 0 and Week 12
  The 25-item Connor-Davidson Resilience Scale (CD-RISC 25) collects information on resilience, which is the ability to thrive despite adversity. The total score ranges from 0 (low resilience) to 100 (higher resilience)

OTHER OUTCOMES:
Tailored physical activity program for elderly African American adults | 1.5 hour focus groups prior to RCT. Recruitment, retention and protocol compliance throughout the intervention
  Use focus groups to gather information needed to tailor a physical activity program

CONTACTS AND LOCATIONS:
Overall Officials: Robert Newton, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwizdala KL, Brouillete R, Beyl R, Johnson W, Hebert C, Carter L, Harris M, Newton RL Jr, Carmichael OT. Exercise Effects on Cognition in Older African Americans: A Pilot Randomized Trial. Front Aging Neurosci. 2022 Jul 22;14:921978. doi: 10.3389/fnagi.2022.921978. eCollection 2022. PMID 35936770
- [Derived] Newton RL Jr, Beyl R, Hebert C, Harris M, Carter L, Gahan W, Carmichael O. A Physical Activity Intervention in Older African Americans: The PAACE Pilot Randomized Controlled Trial. Med Sci Sports Exerc. 2022 Oct 1;54(10):1625-1634. doi: 10.1249/MSS.0000000000002956. Epub 2022 May 7. PMID 35522253